CLINICAL TRIAL: NCT02804373
Title: Effects of Intranasal Administration of Oxytocin in Adults With Prader-Willi Syndrome
Acronym: PRADOTIM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13 6872 03
Record Dates: First submitted 2015-07-10; First posted 2016-06-17 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2020-07

CONDITIONS: Prader-Willi Syndrome
Keywords: oxytocin; adults
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo daily (Placebo Comparator): daily administration of placebo during 28 days : placebo continuous
  Interventions: Drug: Placebo continuous
- 24 IU of oxytocin daily (Active Comparator): 24 IU of daily oxytocin administration during 28 days : oxytocin continuous
  Interventions: Drug: Oxytocin (OXT) continuous
- 24 IU of oxytocin every 3 days (Active Comparator): 24 IU of daily oxytocin every 3 days and placebo the following 2 days after each oxytocin administration during 28 days
  Interventions: Drug: Placebo; Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin (OXT) continuous — Administration of 24 IU of oxytocin daily during 28 days
  Other Names: Syntocinon
  Arms: 24 IU of oxytocin daily
Drug: Placebo — Placebo daily during 28 days
  Arms: 24 IU of oxytocin every 3 days
Drug: Placebo continuous — Placebo administration the following 2 days after each OXT administration, during 28 days.
  Arms: placebo daily
Drug: Oxytocin — Administration of 24 IU of oxytocin every 3 days during 28 days.
  Other Names: Syntocinon
  Arms: 24 IU of oxytocin every 3 days

SUMMARY:
The investigator thinks that the oxytocin (OT) can improve durably and significantly the behavior disorders and thus the socialization but also the satisfaction and could thus be an interesting therapeutic alternative for the patients presenting a Prader-Willi Syndrome (SPW). Although today several studies demonstrated the effects of the OT in various domains of the behavior, the investigator do not know either its specificity of action about the cerebral level, or its duration of action, or the optimal modalities of administration and in particular at patients SPW.

ELIGIBILITY:
Inclusion Criteria:

* Prader-Willi syndrome genetically confirmed
* Absence of extension of the QT interval in the electrocardiogram
* Absence of hypokalemia

Exclusion Criteria:

* Psychiatric troubles
* Anomalies of the heart rhythm in significant ECG
* Hepatic insufficiency
* Renal insufficiency
* Patients presenting a pregnancy or breast-feeding
* High sensibility to OT
* High sensibility to the excipients of the product
* Patients having family history of genetic pathology causing an extension of the interval QT
* Patients having risk factors of advanced twist

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Change in Behaviour as assessed by score variations in specific questionaries | Every day before and after administration of treatment during 28 days
Change in eating Behaviour as assessed by score variations in specific questionaries | Every day before and after administration of treatment during 28 days

SECONDARY OUTCOMES:
Change in eating behaviour as assessed by score variations in hunger visual analogic scale | Every day before and after administration of treatment during 28 days
Cerebral Metabolism variations as assessed by Positron Emission Tomography (PET-scan) | Day 1, day 2 and day 30
  Brain imaging
Cerebral Metabolism variations as assessed by functional Magnetic Resonance Imaging (f-RMI) | Day 1, day 2 and day 29
  Brain imaging
Evaluation of social skills assessed by specific questionnaires | Day 1, day 2 and day 30
Evaluation of executive function assessed by specific questionnaires | Day 1, day 2 and day 30
Evaluation of theory of mind assessed by specific questionnaires | Day 1, day 2 and day 30
Social processing assessed by oculomotor exploration | Day 1, day 2 and day 30
Multisensory processing assessed by Neurovisual task | Day 1, day 2 and day 30
Hormon blood concentration levels as assessed by bioassays | Day 2 and day 30

CONTACTS AND LOCATIONS:
Overall Officials: Maithé TAUBER, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Centre de référence Prader-Willi - Hôpital Purpan, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salles J, Strelnikov K, Carine M, Denise T, Laurier V, Molinas C, Tauber M, Barone P. Deficits in voice and multisensory processing in patients with Prader-Willi syndrome. Neuropsychologia. 2016 May;85:137-47. doi: 10.1016/j.neuropsychologia.2016.03.015. Epub 2016 Mar 16. PMID 26994593